CLINICAL TRIAL: NCT04400630
Title: Functionality and Neurocognition in Patients With Bipolar Disorder After a Physical-exercise Program (FINEXT-BD Study): Protocol of a Randomized Interventionist Program
Brief Title: Functionality and Neurocognition in Patients With Bipolar Disorder After a Physical-exercise Program (FINEXT-BD Study)
Acronym: FINEXT-BD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Principal Investigator, ANA GONZALEZ PINTO, Principal Investigator, Bioaraba Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FINEX-BD
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Longitudinal, interventional, randomized, controlled, simple-blind clinical trial
Who Masked: Investigator
Masking Description: The person in charge of the assessments will not be involved in the treatment program and will be blinded to this process. Study evaluators will be blinded to the treatment branch
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (TAU) (No Intervention): patients without any intervention + treatment as usual (TAU)
- PE intervention+TAU (Experimental): Physical exercise (PE) intervention + treatment as usual (TAU)
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — The experimental group will receive supervised physical exercise treatment by high-intensity interval training (HIT), alternating high and moderate intensities (20 min). The participants will exercise two non-consecutive days per week for 16 weeks under supervision by exercise specialists.
  Arms: PE intervention+TAU

SUMMARY:
This is a study that aimed to deep in the physiopathology of BD and see how, through potential modifiable areas of the patients' lifestyle, the prognosis and evolution of the pathology can be improved.

DETAILED DESCRIPTION:
Randomized interventionist study (ratio 1:1) with two parallel branches, blinded by evaluators (the evaluator does not know the branch of treatment to which the patient belongs )to evaluate if an individualized moderate-to-vigorous physical exercise intensity program as adjuvant therapy to standard drug therapy will improve the functional and neuropsychological status of patients with Bipolar Disorder. The effectiveness of the intervention will be assessed by an extensive battery of clinical tests, physical parameters (e.g. brain structure changes measured by optical coherence tomography) and biological parameters (inflammation, oxidative stress and neurotrophic factors).

The total sample of the study will be 80 patients and a sample of 40 controls (individuals without psychiatric pathology). The sample of patients will be divided into 40 patients in each group at random. In the intervention group, a supervised physical exercise treatment by high-intensity interval training (HIT) will be performed during 16 weeks with 2 sessions per week (32 sessions in total).Three visits will be made in both groups: baseline visit at the beginning of the study, at 4 months (at the end of the intervention) and at 10 months (6 months after the end of the intervention)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bipolar disorder type I according to the criteria of the DSM-5 manual, diagnosis made by structured interview SCID-P.
* The study includes patients with first episode and multiple episodes. At the beginning of the study they must be in euthymia, that is, there will be no current diagnosis of manic, hypomanic or depressive episode. Relapses during follow-up and the presence of subindromial symptoms at any time will not result in exclusion from the study.
* Patients may be treated with any treatment according to clinical guidelines.
* Age: 18-65 years
* Speak Spanish correctly
* Informed consent for the study of the patient

Exclusion Criteria:

* Presence of organic diseases of the central nervous system (CNS) or history of head trauma with loss of consciousness
* Intellectual disability.
* Acute inflammatory disease
* Treatment with anti-inflammatory drugs during the week prior to sample taking
* Pervasive developmental disorders.
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Functionality measured through the scale FAST (4 months) | Change at the end of the training period (4 months)
  The Functioning Assessment Short Test is a brief instrument designed to assess functional impairment in severe mental disorders. The 24 items of the scale cover six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, and leisure time.
Patient Functionality measured through the scale FAST (10 months) | Changes after 10 months
  The Functioning Assessment Short Test is a brief instrument designed to assess functional impairment in severe mental disorders. The 24 items of the scale cover six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, and leisure time.
Patient Functionality measured through the scale GAF (4 months) | Change at the end of the training period (4 months)
  Global Assessment of Functioning (GAF):This scale evaluates with a score from 0 to 100 the level of functioning and the severity of the patient's symptoms, the higher values corresponding to better overall functionality.
Patient Functionality measured through the scale GAF (10 months) | Changes after 10 months
  Global Assessment of Functioning (GAF):This scale evaluates with a score from 0 to 100 the level of functioning and the severity of the patient's symptoms, the higher values corresponding to better overall functionality.
Patient Functionality measured through the Strauss-Carpenter scale (4 months) | Change at the end of the training period (4 months)
  Strauss-Carpenter scale consists of four items rated from 0 to 4 on a Likert-type scale and yields a total score that is calculated by the addition of all item scores: the higher the score, the better is the prognosis.
Patient Functionality measured through the Strauss-Carpenter scale (10) months) | Changes after 10 months
  Strauss-Carpenter scale consists of four items rated from 0 to 4 on a Likert-type scale and yields a total score that is calculated by the addition of all item scores: the higher the score, the better is the prognosis.

SECONDARY OUTCOMES:
TrkB-FL (4 months) | Change at the end of the training period (4 months)
  Expression of BDNF: TrkB-FL
TrkB-FL (10 months) | Changes after 10 months
  Expression of BDNF: TrkB-FL
TrkB-T (4 months) | Change at the end of the training period (4 months)
  Expression of BDNF:TrkB-T
TrkB-T (10 months) | Changes after 10 months
  Expression of BDNF:TrkB-T
BDNF (4 months) | Change at the end of the training period (4 months)
  Peripheral BDNF levels
BDNF (10 months) | Changes after 10 months
  Peripheral BDNF levels
Presence of depressive symptoms (4 months) | Change at the end of the training period (4 months)
  Hamilton Depression Scale (HDRS-21)
Presence of depressive symptoms (10 months) | Changes after 10 months
  Hamilton Depression Scale (HDRS-21)
VO2Peak in CPET (4 months) | Change at the end of the training period (4 months)
  Value of VO2Peak (L min-1) in cardiopulmonary exercise test (CPET)
VO2Peak in CPET (10 months) | Changes after 10 months
  Value of VO2Peak (L min-1) in cardiopulmonary exercise test (CPET)
Relative VO2Peak in CPET (4 months) | Change at the end of the training period (4 months)
  Value of relative VO2Peak (mL kg-1 min-1) in cardiopulmonary exercise test (CPET)
Relative VO2Peak in CPET (10 months) | Changes after 10 months
  Value of relative VO2Peak (mL kg-1 min-1) in cardiopulmonary exercise test (CPET)
METs in CPET (4 months) | Change at the end of the training period (4 months)
  Value of metabolic equivalents in cardiopulmonary exercise test (CPET)
METs in CPET (10 months) | Changes after 10 months
  Value of metabolic equivalents in cardiopulmonary exercise test (CPET)
VT1 and VT2 in CPET (4 months) | Change at the end of the training period (4 months)
  Value of first and second ventilatory threshold (VT1 and VT2)(mL kg-1 min-1) metabolic equivalents in cardiopulmonary exercise test (CPET)
VT1 and VT2 in CPET(10 months) | Changes after 10 months
  Value of first and second ventilatory threshold (VT1 and VT2)(mL kg-1 min-1) metabolic equivalents in cardiopulmonary exercise test (CPET)
HRpeak in CPET (4 months) | Change at the end of the training period (4 months)
  Value of HRpeak in cardiopulmonary exercise test (CPET)
HRpeak in CPET (10 months) | Changes after 10 months
  Value of HRpeak in cardiopulmonary exercise test (CPET)
OCT Study of the retina by optical tomography (4 months) | Change at the end of the training period (4 months)
  RFNL, GCL and IPL thickness in the two eyes, with each layer divided into segments: overall, temporal, nasal, superior and inferior.
OCT Study of the retina by optical (10 months) | Changes after 10 months
  RFNL, GCL and IPL thickness in the two eyes, with each layer divided into segments: overall, temporal, nasal, superior and inferior.
Muscle mass (4 months) | Change at the end of the training period (4 months)
  Anthropometric measures muscle mass (g)
Muscle mass (10 months) | Changes after 10 months
  Anthropometric measures muscle mass (g)
Fat mass (%)(4 months) | Change at the end of the training period (4 months)
  Anthropometric measures Fat mass (%)
Fat mass (%) (10 months) | Changes after 10 months
  Anthropometric measures Fat mass (%)
Bone mineral content (4 months) | Change at the end of the training period (4 months)
  Anthropometric measures: Bone mineral density (g/cm^2) shall be determined by Dual Energy X-Ray Absorptiometry (DXA).
Bone mineral content (4 months) | Changes after 10 months
  Anthropometric measures: Bone mineral density (g/cm^2) shall be determined by Dual Energy X-Ray Absorptiometry (DXA).
Appendicular muscle mass (4months) | Change at the end of the training period (4 months)
  Anthropometric measures: appendicular muscle mass (g) will also be determined by adding up the muscle mass of both arms and legs.
Appendicular muscle mass (10 months) | Changes after 10 months
  Anthropometric measures: appendicular muscle mass (g) will also be determined by adding up the muscle mass of both arms and legs.
Oxidative stress (4 months) | Change at the end of the training period (4 months)
  Oxidative stress: Total Antioxidant Status (TAS), Glutathione peroxidase (GPx) y - Glutathione (GSH), Lipid Peroxidation (TBARS) y Nitrite (NO2)
Oxidative stress (10 months) | Changes after 10 months
  Oxidative stress: Total Antioxidant Status (TAS), Glutathione peroxidase (GPx) y - Glutathione (GSH), Lipid Peroxidation (TBARS) y Nitrite (NO2)
Inflammation (4 months) | Change at the end of the training period (4 months)
  Cytokine levels: IL6 and prostaglandin Levels PGE2
Inflammation (10 months) | Changes after 10 months
  Cytokine levels: IL6 and prostaglandin Levels PGE2
Manic symptoms using the (YMRS) (4 months) | Change at the end of the training period (4 months)
  Young Mania Rating Scale (YMRS): The total score ranges from 0-60, with the status of euthymia being classified as getting 6 or fewer points, hypomania as getting 12 or more points, and mania as getting between 20 and 60 points.
Manic symptoms using the (YMRS) (10 months) | Changes after 10 months
  Young Mania Rating Scale (YMRS): The total score ranges from 0-60, with the status of euthymia being classified as getting 6 or fewer points, hypomania as getting 12 or more points, and mania as getting between 20 and 60 points.
Body mass (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Body mass (kg)
Body mass (10 months) | Changes after 10 months
  Physical parameters: Body mass (kg)
Height (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Height (cm)
Height (10 months) | Changes after 10 months
  Physical parameters: Height (cm)
BMI (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Body mass index (kg/m2)
BMI (10 months) | Changes after 10 months
  Physical parameters: Body mass index (kg/m2)
Waist circumference (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Waist circumference (cm)
Waist circumference (4 months) | Changes after 10 months
  Physical parameters: Waist circumference (cm)
SBP and DBP (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Systolic and diastolic blood pressure (mm Hg) measured taken from the right arm in a seated and relaxed position by using a life-support monitor
SBP and DBP (10 months) | Changes after 10 months
  Physical parameters: Systolic and diastolic blood pressure (mm Hg) measured taken from the right arm in a seated and relaxed position by using a life-support monitor
TG (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Serum levels of triglycerides (mg/dl )
TG (10 months) | Changes after 10 months
  Physical parameters: Serum levels of triglycerides (mg/dl )
Glucose (4 months) | Change at the end of the training period (4 months)
  Physical parameters: Glucose (mg/dl)
Glucose (10 months) | Changes after 10 months
  Physical parameters: Glucose (mg/dl)
HDL (4 months) | Change at the end of the training period (4 months)
  Physical parameters: HDL colesterol (mg/dl)
HDL (10 months) | Changes after 10 months
  Physical parameters: HDL colesterol (mg/dl)
Patient symptom severity measured through the scale CGI (4 months) | Change at the end of the training period (4 months)
  The Clinical Global Impression Scale (CGI): consists of two subscales. Each subscale has a single item scored between 0, not evaluated, to 7 which corresponds to the maximum severity (severity subscale) or to a state of no improvement and aggravated worsening of the symptomatology (improvement subscale).
Patient symptom severity measured through the scale CGI (10 months) | Changes after 10 months
  The Clinical Global Impression Scale (CGI): consists of two subscales. Each subscale has a single item scored between 0, not evaluated, to 7 which corresponds to the maximum severity (severity subscale) or to a state of no improvement and aggravated worsening of the symptomatology (improvement subscale).
Cognitive functioning measured through CVLT (10 months) | Changes after 10 months
  California Verbal Learning Test
Cognitive functioning measured through CVLT (4 months) | Change at the end of the training period (4 months)
  California Verbal Learning Test
Cognitive functioning measured through WSCT (10 months) | Changes after 10 months
  Computerized version of Wisconsin Card Sorting Test: This test consists of cards depicting simple geometric figures that vary in color, shape, and number. Examinees must sort cards in accordance with one of three viable rules, i.e., according to the color, shape, or number of the depicted objects
Cognitive functioning measured through WSCT (4 months) | Change at the end of the training period (4 months)
  Computerized version of Wisconsin Card Sorting Test: This test consists of cards depicting simple geometric figures that vary in color, shape, and number. Examinees must sort cards in accordance with one of three viable rules, i.e., according to the color, shape, or number of the depicted objects
Cognitive functioning measured through (SCWT) (10 months) | Changes after 10 months
  The Stroop Color and Word Test: Individuals are required to read three different tables as fast as possible. Two of them represent the "congruous condition" in which participants are required to read names of colors (color-words) printed in black ink (W) and name different color patches (C). Conversely, in the third table, named color-word (CW) condition, color-words are printed in an inconsistent color ink.
Cognitive functioning measured through (SCWT) (4 months) | Change at the end of the training period (4 months)
  The Stroop Color and Word Test: Individuals are required to read three different tables as fast as possible. Two of them represent the "congruous condition" in which participants are required to read names of colors (color-words) printed in black ink (W) and name different color patches (C). Conversely, in the third table, named color-word (CW) condition, color-words are printed in an inconsistent color ink.

CONTACTS AND LOCATIONS:
Overall Officials: Ana María Gonzalez-Pinto, Principal Investigator — BIOARABA HRI
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Alava, Spain

REFERENCES:
- [Derived] Garcia S, Gorostegi-Anduaga I, Garcia-Corres E, Maldonado-Martin S, MacDowell KS, Bermudez-Ampudia C, Apodaca MJ, Perez-Landaluce I, Tobalina-Larrea I, Leza JC, Gonzalez-Pinto A. Functionality and Neurocognition in Patients With Bipolar Disorder After a Physical-Exercise Program (FINEXT-BD Study): Protocol of a Randomized Interventionist Program. Front Psychiatry. 2020 Oct 29;11:568455. doi: 10.3389/fpsyt.2020.568455. eCollection 2020. PMID 33240125